CLINICAL TRIAL: NCT04534348
Title: Study on the Reduction of Catheter-related Infections by Use of Self-disinfecting Venous and Arterial Access Caps
Acronym: STERILE
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Maria J.G.T. Vehreschild, Prof. MD, University of Cologne
Other Study IDs: STERILE
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: CLABSI - Central Line Associated Bloodstream Infection; Catheter-Related Blood Stream Infection
Keywords: CLABSI; CRBSI; Blood Stream Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control: All central-line-associated blood stream infections (CLABSI) diagnosed during the year previous the implementation of 70% isopropyl alcohol-impregnated Curos catheter caps
- CUROS: All central-line-associated blood stream infections (CLABSI) diagnosed during the year after the implementation of 70% isopropyl alcohol-impregnated Curos catheter caps
  Interventions: Device: 70% isopropyl alcohol-impregnated catheter caps

INTERVENTIONS:
Device: 70% isopropyl alcohol-impregnated catheter caps — Implementation of 70% isopropyl alcohol-impregnated catheter caps in order to assess the number of CLABSI diagnosed during 1 Year
  Other Names: CUROS (3M); self disinfecting catheter caps
  Groups: CUROS

SUMMARY:
Observational study on the reduction of catheter-related Infections by use of self-disinfecting venous and arterial access caps (Curos caps ;3M, Saint Paul, MN, USA)

ELIGIBILITY:
Inclusion Criteria:

* every patient in the hemato-oncological department who received at least one CVC was included in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in the hemato-oncological department at the University Clinic in Cologne, Germany, receiving a central-line catheter during one year previous to the implementation of alcohol-impregnated catheter caps as well as all patients receiving a central-line catheter during the 12 months following the implementation of CUROS were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Number of CLABSI | 12 Months
  To assess the clinical efficacy of Curos in preventing CLABSI in a high-risk department (oncology and ICU)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No